Evaluation of Acuvue Oasys 1-Day contact lenses in new wearers

Protocol CR-6565

Version: 2.0

Date: 12 March 2024

Investigational Products: ACUVUE OASYS® 1-DAY with HydraLuxe™ TECHNOLOGY

Keywords: R&D Sphere, New Wearer, senofilcon A marketed product (ACUVUE OASYS® 1-DAY with HydraLuxe<sup>TM</sup> TECHNOLOGY), Daily Wear, Daily Disposable, dispensing, Eye-Cept preservative free rewetting drops, refraction, Insertion and Removal training, neophytes, confidence survey, motivation survey, CLUE comfort, CLUE vision, CLUE handling.

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This clinical trial will be conducted in compliance with ISO 14155:2020 Clinical investigation of medical devices for human subjects – Good clinical practice<sup>1</sup>, and the Declaration of Helsinki.<sup>2</sup>

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

# TABLE OF CONTENTS

| P | ROT | OCOL TITLE, NUMBER, VERSION AND DATE | 6 |
|---|---|---|---|
| S | PON | SOR NAME AND ADDRESS | 6 |
| M | EDI | CAL MONITOR | 6 |
| A | UTH | ORIZED SIGNATURES | 7 |
| C | HAN | IGE HISTORY | 8 |
| S | YNO | PSIS | 9 |
| C | OMN | MONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS | 13 |
| 1. | I | NTRODUCTION AND BACKGROUND | 14 |
| | 1.1. | Name and Descriptions of Investigational Products | 14 |
| | 1.2. | Intended Use of Investigational Products | 14 |
| | 1.3. | Summary of Findings from Nonclinical Studies | 14 |
| | 1.4. | Summary of Known Risks and Benefits to Human Subjects | 14 |
| | 1.5. | Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study | 14 |
| 2. | 5 | STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 15 |
| | 2.1. | Objectives | 15 |
| | 2.2. | Endpoints | 15 |
| | 2.3. | Hypotheses | 16 |
| 3. | | FARGETED STUDY POPULATION | 16 |
| | 3.1. | General Characteristics | 16 |
| | 3.2. | Inclusion Criteria | 16 |
| | 3.3. | Exclusion Criteria | 17 |
| | 3.4. | Enrollment Strategy | 17 |
| 4. | 5 | STUDY DESIGN AND RATIONALE | 17 |
| | 4.1. | Description of Study Design | 17 |
| | 4.2. | Study Design Rationale | 17 |
| | 4.3. | Enrollment Target and Study Duration | 18 |
| 5. | 7 | TEST ARTICLE ALLOCATION AND MASKING | 18 |
| | 5.1. | Test Article Allocation | 18 |
| | 5.2. | Masking | 18 |
| | 5.3. | Procedures for Maintaining and Breaking the Masking | 18 |
| 6. | 5 | STUDY INTERVENTION | 18 |
| | 6.1. | Identity of Test Articles | 18 |
| | 6.2. | Ancillary Supplies/Products | 19 |
| | 6.3. | Administration of Test Articles | 19 |
| | 6.4. | Packaging and Labeling | 19 |
| | 6.5. | Storage Conditions | 20 |
| | 6.6. | Collection and Storage of Samples | 20 |
| | 6.7. | Accountability of Test Articles | 20 |

| 7. | STU | JDY EVALUATIONS | 20 |
|---|---|---|---|
| | 7.1. | Time and Event Schedule | 20 |
| | 7.2. | Detailed Study Procedures | 22 |
| | VIS | IT 1 | 22 |
| | VIS | IT 2 | 30 |
| | VIS | IT 3 | 33 |
| | FIN | AL EVALUATION | 34 |
| | 7.3. | Unscheduled Visits | 35 |
| | 7.4. | Laboratory Procedures | 36 |
| 8. | SUI | BJECTS COMPLETION/WITHDRAWAL | 36 |
| | 8.1. | Completion Criteria | 36 |
| | 8.2. | Withdrawal/Discontinuation from the Study | 36 |
| 9. | PRE | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 37 |
| | 9.1. | Systemic Medications | 37 |
| 10. | DE | VIATIONS FROM THE PROTOCOL | 37 |
| 11. | STU | JDY TERMINATION | 38 |
| 12. | PRO | OCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 39 |
| 13. | AD | VERSE EVENTS | 40 |
| | 13.1. | Definitions and Classifications | 40 |
| | 13.2. | Assessing Adverse Events | 41 |
| | 13.2 | 2.1. Causality Assessment | 42 |
| | 13.2 | 2.2. Severity Assessment | 42 |
| | 13.3. | Documentation and Follow-Up of Adverse Events | 42 |
| | 13.4. | Reporting Adverse Events | 43 |
| | 13.4 | 1. Reporting Adverse Events to Sponsor | 43 |
| | 13.4 | 2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities | 44 |
| | 13.5. | Event of Special Interest | 44 |
| | 13.6. | Reporting of Pregnancy | 44 |
| 14. | STA | ATISTICAL METHODS | 44 |
| | 14.1. | General Considerations | 44 |
| | 14.2. | Sample Size Justification | 45 |
| | 14.3. | Analysis Populations | 45 |
| | 14.4. | Level of Statistical Significance. | 45 |
| | 14.5. | Primary Analysis | 45 |
| | 14.6. | Secondary Analysis | 45 |
| | 14.7. | Exploratory Analysis | 45 |
| | 14.8. | Interim Analysis | 46 |
| | 14.9. | Procedure for Handling Missing Data and Drop-Outs | 46 |
| | 14.10. | Procedure for Reporting Deviations from Statistical Plan | 46 |

| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 46 |
|---|---|---|---|
| | 15.1. | Electronic Case Report Form/Data Collection | 46 |
| | 15.2. | Subject Record | 46 |
| | 15.3. | Trial Registration on ClinicalTrials.gov | 47 |
| 16. | DA | TA MANAGEMENT | 47 |
| | 16.1. | Access to Source Data/Document | 47 |
| | 16.2. | Confidentiality of Information | 47 |
| | 16.3. | Data Quality Assurance | 47 |
| | 16.4. | Data Monitoring Committee (DMC) | 47 |
| 17. | CL | NICAL MONITORING | 48 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | 48 |
| | 18.1. | Study-Specific Design Considerations | 48 |
| | 18.2. | Investigator Responsibility | 48 |
| | 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 48 |
| | 18.4. | Informed Consent | 49 |
| | 18.5. | Privacy of Personal Data | 50 |
| 19. | STU | JDY RECORD RETENTION | 51 |
| 20. | FIN | IANCIAL CONSIDERATIONS | 51 |
| 21. | PU | BLICATION | 51 |
| 22. | RE | FERENCES | 51 |
| AP | PEND | IX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 53 |
| AP | PEND | IX B: PATIENT INSTRUCTION GUIDE | 64 |
| AP | PEND | IX C: PACKAGE INSERT (APPROVED PRODUCT) | |
| AP | PEND | IX D: | 94 |
| | | LENS FITTING CHARACTERISTICS | |
| | | SUBJECT REPORTED OCULAR SYMPTOMS | 101 |
| | | FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE | 103 |
| | | DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIVE ERROR | 108 |
| | | BIOMICROSCOPY SCALE | 114 |
| | | DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION | 120 |
| | | PATIENT REPORTED OUTCOMES | 125 |
| | | WHITE LIGHT LENS SURFACE WETTABILITY | 127 |
| AP | PEND | IX E: WORK AID: INSERTION AND REMOVAL TRAINING GUIDE | 129 |
| AP | PEND | IX F: GUIDELINES FOR COVID-19 RISK MITIGATION | 139 |
| PR | OTOC | OL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 150 |
| | | F TABLES | 10 |
| | | Fest Articles | |
| 1 a | oie 2: <i>I</i> | Ancillary Supplies | 19 |

| Table 3: Time and Events | 21 |
|----------------------------------------------------------|----|
| Table 4: Disallowed systemic medications | 37 |
| Table 5: Examples of major and minor protocol deviations | 38 |
| LIST OF FIGURES | |
| Figure 1: Study Flowchart | 12 |

## PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Evaluation of Acuvue Oasys 1-Day contact lenses in new wearers

Protocol Number: CR-6565

Version: 2.0

Date: 12 March 2024

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### AUTHORIZED SIGNATURES

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, <sup>3</sup> ISO 14155:2020, <sup>1</sup> and the Declaration of Helsinki. <sup>2</sup>

| Author & Study | | |
|------------------------|---------------------------------|-------------|
| Responsible Clinician | See Electronic Signature Report | |
| | | DATE |
| | _ | |
| Medical Monitor | See Electronic Signature Report | |
| | | DATE |
| eranna abw | * | |
| Clinical Operations | Cas Electronia Cionatura Banaut | |
| Manager | See Electronic Signature Report | DATE |
| Biostatistician | San Electronic Signature Bonart | |
| Biostatistician | See Electronic Signature Report | DATE |
| Biostatistician | | |
| Reviewer | See Electronic Signature Report | |
| | | DATE |
| Data Management | | |
| | See Electronic Signature Report | DATE |
| M 1 10 C+ 000 | C. Fl. C. C. D. | <del></del> |
| Medical Safety Officer | See Electronic Signature Report | DATE |
| A CONTRACTOR | C. Fl. C. C. D. D. | |
| Approver | See Electronic Signature Report | DATE |

# **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and<br>Section Number(s) Affected | Justification<br>for Change | Date |
|---|---|---|---|---|
| 1.0 | | Original Protocol | N/A | 23 Feb 2024 |
| 2.0 | | Updated the primary objective in section 1.2 to match the other sections of the protocol. | | 12MAR2024 |

## **SYNOPSIS**

| Protocol Title | Evaluation of Acuvue Oasys 1-Day contact lenses in new wearers |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Clinical trial phase: |
| | Post Market |
| | Design control phase: Post-Marketing, Phase 4 |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the Sponsor. |
| Test Article: | Approved Product: ACUVUE OASYS® 1-DAY with HydraLuxe <sup>TM</sup> |
| | TECHNOLOGY (AO1D) |
| Wear and Replacement | Wear Schedule: Daily wear (DW) |
| Schedules | Replacement Schedule: Daily disposable (DD) |
| Objectives | <b>Primary Objective:</b> The primary objective of this study is to estimate the |
| | incidence rate (percentage) of eyes with clinically significant slit-lamp findings (Grade 3 or 4) related to the study lens after approximately 2-weeks |
| | of lens wear. |
| | Exploratory Objectives: The other objectives are to measure commitment |
| | to lens wear in neophyte subjects after approximately two weeks of wearing |
| | experience, measure Insertion & Removal (I&R) skills, evaluate new wearer |
| | confidence and motivation for lens wear, and assess lens performance (CLUE vision, comfort & handling scores). |
| Study Endpoints | Primary Endpoints: |
| Study Enapoints | 1. Incidence (percentage) of eyes with Grade 3 or 4 slit lamp findings |
| | related to the study lenses after 2-week of lens wear. |
| | Exploratory Endpoints: |
| | • Commitment to lens wear: Do you want to continue to wear |
| | contact lenses after this study? (Yes or No) |
| | <ul> <li>Reason for discontinuation (if applicable).</li> <li>Time for lens insertion OU</li> </ul> |
| | Time for lens insertion OU Time for lens removal OU |
| | New wearer confidence level |
| | New wearer motivation level |
| | Lens performance (CLUE vision, comfort, handling scores) |
| Study Design | This is a multi-site, bilateral, dispensing, non-randomized, uncontrolled, |
| | unmasked, single arm study. Each subject will be fitted with the study lenses |
| | and dispensed for approximately 14 days of wear. |
| | There will be a total of 3 visits: |
| | Visit 1: Screening, baseline evaluation and lens fitting. Dispense for $7 \pm 1$ |
| | days. |
| | Visit 2: Follow up #1; Dispense an additional supply for $7 \pm 1$ days. |
| | Visit 3: Follow up #2; Final evaluation. |
| | See the flow chart at the end of the synopsis table for the schematic of the |
| | study visits and procedures of main observations (Figure 1). |
| Sample Size | Approximately 40 neophyte subjects will be enrolled into the study. It is |
| * | anticipated that approximately 30 subjects will complete the study. |
| Study Duration | The study enrollment period is approximately 8 weeks. Once enrolled, |
| | subjects will be in the study for about 2 weeks, making the total study duration |
| | about 10 weeks from the first subject first visit (FSFV) to last subject last visit (LSLV). |
| | (LSLY). |

| Anticipated Study Population | Healthy pediatric and adult subjects, ages 13 to 39 (inclusive), of any race or |
|---|---|
| Anticipated Study Population | |
| | ethnicity that have never trialed or placed lenses on eye (neophytes), that meet |
| E1: 11:12- C : 1 1- : | the eligibility criteria for the study. |
| Eligibility Criteria - Inclusion | Potential subjects must satisfy all of the following criteria to be enrolled in the |
| | study: |
| | Inclusion Criteria following Screening |
| | The subject must: |
| | 1. Read, understand, and sign the Statement of Informed Consent and |
| | receive a fully executed copy of the form. (For subjects aged 18 and |
| | older) |
| | 2. Read (or be read to) and sign the Children's Assent (Information and |
| | Assent Form) and receive a fully executed copy of the form. (For |
| | subjects aged 13 to 17) |
| | 3. Have parents or legal guardians who must read, understand, and sign |
| | the Statement of Informed Consent (Parental Permission Form and |
| | Authorization to Use and Disclose Medical Information). (For |
| | subjects aged 13 to 17) |
| | 4. Appear able and willing to adhere to the instructions set forth in this |
| | clinical protocol. |
| | 5. Be between 13 and 39 (inclusive) years of age at the time of |
| | screening. |
| | 6. By self-report, having never worn any type of contact lenses and |
| | never attempted to insert contact lenses. |
| | 7. Have a pair of prescription glasses on hand that corrects distance |
| | vision, if determined to be required by the investigator. |
| | Inclusion Criteria at Baseline Evaluation |
| | 8. The magnitude of the cylindrical component of the subject's vertex- |
| | corrected distance refraction must be $\leq 0.75$ DC in each eye. |
| | 9. Subject must have a vertex corrected distance sphero-cylindrical |
| | refraction in the range such that appropriate spherical lens powers |
| | are available for correction in both eyes. The spherical lens powers |
| | available in this study are: |
| | a1.00 to -6.00 (in 0.25D steps) |
| | 10. Best corrected monocular distance visual acuity must be 20/20 <sup>-3</sup> or |
| | better in each eye. |
| Eligibility Criteria – | Potential subjects who meet any of the following criteria will be excluded |
| Exclusion | from participating in the study: |
| | Exclusion Criteria following Screening |
| | The subject must not: |
| | 1. Be currently pregnant or lactating. |
| | 2. Be currently using any ocular medications or have any ocular |
| | infection of any type. |
| | 3. By self-report, have any ocular or systemic disease, allergies, or |
| | infection, or use medications that the investigator believes might |
| | contraindicate or interfere with contact lens wear, or otherwise |
| | compromise the study endpoints. See section 9.1 for additional |
| | details regarding systemic medications. |
| | 4. Have previously participated in a contact lens, contact lens primary |
| | package, or lens care related clinical trial. |
| | 5. Be an employee (e.g., Investigator, Coordinator, Technician) or |
| | immediate family member of an employee (including partner, child, |
| | parent, grandparent, grandchild, or sibling of the employee or their |
| | spouse) of the clinical site. |
| l- | . / |

| | Exclusion Criteria at Baseline Evaluation The subject must not: 6. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings or other corneal, eyelid, or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including significant blepharitis, entropion, ectropion, ptosis, chalazia, recurrent styes, pterygium, significant dry eye disease, history of recurrent corneal erosions, aphakia, corneal distortion, herpetic keratitis). 7. Have a history of strabismus or amblyopia. 8. Have fluctuations in vision due to clinically significant dry eye or other ocular or systemic conditions. 9. Have had or have planned (within the study period) any ocular or intraocular surgery or procedures (e.g., PRK, LASIK, IPL, blepharoplasty, etc.) |
|---|---|
| Disallowed | See section 9.1 for details regarding disallowed systemic medications. |
| Medications/Interventions | |
| Measurements and | The key procedures associated with this study will be: |
| Procedures | Refraction |
| | Evaluation and grading of ocular physiology using a slit lamp |
| | biomicroscope. |
| | Contact lens I&R training. L&B skills measurement (a.g., time to insertion) |
| | <ul><li>I&amp;R skills measurement (e.g., time to insertion).</li><li>Contact lens fitting.</li></ul> |
| | <ul> <li>Evaluation of subjective comfort, vision and handling using the CLUE questionnaire.</li> </ul> |
| | Evaluation of subject's confidence and motivation for lens wear (survey). |
| Microbiology or Other | None. |
| Laboratory Testing | |
| Study Termination | The occurrence of an Unanticipated Adverse Device Effect (UADE) or Serious Adverse Event (SAE) for which a causal relationship to a test article cannot be ruled out, could result in stopping further dispensing of the marketed product. In the event of a UADE or SAE, the Sponsor Medical Monitor may review the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | BioTrue Multipurpose contact lens solution, LacriPure, Eye-Cept, or another preservative free rewetting drop. Sodium Fluorescein. |
| | Supply the subject a bottle of contact lens solution for rinsing purposes, if necessary. |
| Principal Investigator(s) and<br>Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |
| | This study will utilize approximately 5 clinical sites. |

Figure 1: Study Flowchart

### Visit 1: Screening

Statement of Informed Consent, Childrens Assent (if applicable)

Demographics

Medical History & Concomitant Medications

Eligibility after Screening

#### Visit 1: Baseline Evaluation

Subject Reported Ocular Symptoms

Baseline confidence & motivation questionnaire

Baseline (entrance) visual acuity

Spherocylindrical Refraction and Distance VA

Slit Lamp Biomicroscopy

Eligibility at Baseline

#### Visit 1: Lens Fitting

Lens power selection

I&R training (staff trains the subject)

I&R learning session (timed)

Lens fit assessment

Spherical over-refraction, Modification (if applicable)

Subject Reported Ocular Symptoms

Patient reported outcomes (Post fit questionnaire)

Patient education and instructions

Dispense 7± 1 days

#### Visit 2: Follow up #1

Wear compliance

Subject Reported Ocular Symptoms

Confidence & Motivation Questionnaire

Patient reported outcomes (Post fit questionnaire)

Removal of lenses (timed)

Slit Lamp Biomicroscopy

Insertion of lenses (timed)

Lens fit assessment

Continuance & Dispense 7± 1 days

## Visit 3: Follow up #2

Wear compliance

Subject Reported Ocular Symptoms

Confidence & Motivation Questionnaire

Patient reported outcomes (Post fit questionnaire)

Removal of lenses, re-insertion of lenses (timed)

Lens fit assessment

Slit Lamp Biomicroscopy

#### **Final Evaluation**

Commitment to lens wear questionnaire

#### COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADE Adverse Device Effect

ADHD Attention Deficit Hyperactivity Disorder AE Adverse Event/Adverse Experience

AO1D ACUVUE OASYS® 1-DAY with HydraLuxe™ TECHNOLOGY

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

D Diopter

DMC Data Monitoring Committee
eCRF Electronic Case Report Form
EDC Electronic Data Capture
FDA Food and Drug Administration
GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

HL Hand Length

HVID Horizontal Visible Iris Diameter

IB Investigator's Brochure

ICH The International Council for Harmonization

IEC Independent Ethics Committee
IRB Institutional Review Board
I&R Insertion and Removal

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc. LASIK Laser-Assisted in Situ Keratomileusis

OD Right Eye
OS Left Eye
OU Both Eyes

MPMVA Maximum Plus to Maximum Visual Acuity

PAH Palpebral aperture height
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

PW Palm Width QA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan
SAS Statistical Analysis System
SD Standard Deviation

UADE Unanticipated Adverse Device Effect
USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

#### 1.1. Name and Descriptions of Investigational Products

This study will use the commercially available spherical ACUVUE OASYS® 1-DAY with HydraLuxe<sup>TM</sup> TECHNOLOGY (AO1D) contact lenses. Further details about the Test article are found in section 6 of this protocol.

#### 1.2. Intended Use of Investigational Products

The intended use of the study lenses is for correcting myopia. There will be one treatment in this study. During the study, subjects will wear AO1D lenses bilaterally in daily wear, daily disposable modality over the course of approximately two weeks. Since the primary objective of this study is to estimate the incidence rate (percentage) of eyes with clinically significant slit-lamp findings (Grade 3 or 4) related to the study lens after approximately 2-weeks of lens wear, subjects will not be required to adhere to any specific minimum lens wear requirements, however, they will be instructed to only wear the lenses during waking hours and educated on typical wear time (e.g., maximum 14-16 hours per day).

#### 1.3. Summary of Findings from Nonclinical Studies

Not Applicable – Marketed product only.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The following risks/adverse events and clinical benefits can be associated with wearing soft contact lenses in general:

- The eyes may burn, sting and/or itch.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers, and corneal erosion.
- There may be the potential for other physiological observations, such as local or generalized edema,
- corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also
  occur.
- Soft contact lenses, like spectacle lenses, provide correction of refractive error.

For the most comprehensive risk and benefit information regarding study lenses refer to the package insert of the marketed product (Appendix C).

#### 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Recent review of the literature points to several factors that may contribute to new wearer dropout. Sulley *et al* found that the main reasons for discontinuation were problems with vision (41%), discomfort (36%), and handling problems  $(25\%)^4$ .

This study will measure commitment to lens wear in a healthy neophyte population. Eligible subjects will be trained and fitted into a commercially available daily disposable contact lens brand (AO1D), known for its acceptable clinical performance. After approximately two weeks of wear experience, subjects will be interviewed about their commitment to lens wear. Subjects may drop out of the study prematurely, and if so, the reason for dropping out will be documented.

For the most comprehensive information regarding study lenses refer to the package insert of the marketed product (Appendix C).

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

<u>Primary Objective:</u> The primary objective of this study is to estimate the incidence rate (percentage) of eyes with clinically significant slit-lamp findings (Grade 3 or 4) related to the study lens after approximately 2-weeks of lens wear.

<u>Exploratory Objectives:</u> The other objectives are to measure commitment to lens wear in neophyte subjects after approximately two weeks of wearing experience, measure Insertion & Removal (I&R) skills, evaluate new wearer confidence and motivation for lens wear, and assess lens performance (CLUE vision, comfort & handling scores).

#### 2.2. Endpoints

#### **Primary Endpoint:**

### 1. Percentage of eyes with slit-lamp findings (Grade 3 or 4) related to study lens wear:

Slit Lamp Findings (Grade 3 or higher) will be assessed for each subject eye at all study visits (scheduled and unscheduled). However, the primary endpoint will be the percentage of eyes with Grade 3 or higher SLFs related to study lens wear, after approximately 2 weeks of lens wear. SLFs will be evaluated and classified using the FDA Grading scale rating from 0 to 4, where Grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e., Grade 1=trace, Grade 2= mild, Grade 3=moderate and Grade 4= severe).

#### **Other Exploratory Endpoints:**

- 1. **Commitment to lens wear:** Do you want to continue to wear contact lenses after this study? (Response set: Yes, No)
- 2. **Reasons for Discontinuation** (if applicable): Which of the following is the main reason why you want to **stop** wearing contact lenses? (Response set: They were uncomfortable to wear, My eyes were too dry to wear them, I didn't like my vision with contacts, They were too difficult to put on and take off, They were more trouble than it's worth, I'm concerned about the cost, and Other reason [free text])

#### 3. **Insertion Time:**

Insertion time is quantified as the total time (in minutes and seconds) it takes for the subject to <u>insert both lenses</u> (OU). Insertion time will be collected at the initial fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear. The insertion time is a continuous endpoint.

#### 4. Removal Time:

Removal time is quantified as the total time (in minutes and seconds) it takes for the subject to <u>remove</u> their lenses (OU) at three different time points – at the initial fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear. The removal time is a continuous endpoint.

#### 5. Confidence:

New wearer **confidence** (**for lens wear**) will be assessed at baseline (prior to lens fitting), post fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear using the individual questionnaire item: How confident do you feel in your ability to successfully **put on** contact lenses? (Response Set: Not confident, A little confident, Somewhat confident, Confident, Highly confident). (Response Set: No confidence/Little Confidence/Some Confidence/Confident/High Confidence). New wearer confidence is an ordinal categorical endpoint.

#### 6. Motivation:

New wearer motivation (for lens wear) will be assessed at baseline (prior to lens fitting), post lens fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear using the individual questionnaire item: How motivated are you to wear contact lenses? (Response Set: I am not

motivated, /I am a little motivated, /I am somewhat motivated, /I am motivated, /I am highly motivated). New wearer motivation is an ordinal categorical endpoint.

7. **CLUE Vision, Comfort, and Handling scores** will be collected at the initial fitting, after approximately 1-week of wear, and after approximately 2 weeks of wear. The CLUE vision, comfort and handling scores are continuous endpoints.

Subjective comfort, vision, handling scores will be assessed using the Contact Lens Use Experience (CLUE<sup>TM</sup>)<sup>5</sup> questionnaire after approximately 30 minutes of lens wear (post initial fitting), and after approximately 1 and 2 weeks of wear. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.

### 2.3. Hypotheses

Not applicable. All study endpoints will be summarized descriptively.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Subjects will be healthy male and female volunteers of any race and ethnicity that meet the inclusion and exclusion criteria. Subjects who are eligible to be enrolled will be between the ages of 13 and 39 years old. Subjects younger than 18 years old are considered minors and will be required to be accompanied by a parent or a legal guardian. Appropriate Informed Consent forms and Children's Assent forms will be presented, and ample time will be provided for the subjects and their parent or legal guardian to ask questions and make an informed decision.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

#### **Inclusion Criteria following Screening**

The subject must:

- 1. Read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form (For subjects aged 18 and older)
- 2. Read (or be read to) and sign the Children's Assent (Information and Assent Form) and receive a fully executed copy of the form. (For subjects aged 13 to 17)
- 3. Have parents or legal guardians who must read, understand, and sign the Statement of Informed Consent (Parental Permission Form and Authorization to Use and Disclose Medical Information). (For subjects aged 13 to 17)
- 4. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 5. Be between 13 and 39 (inclusive) years of age at the time of screening.
- 6. By self-report, having never worn any type of contact lenses and never attempted to insert contact lenses.
- 7. Have a pair of prescription glasses on hand that corrects distance vision, if determined to be required by the investigator.

#### **Inclusion Criteria at Baseline Evaluation**

- 8. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be  $\leq 0.75$  DC in each eye.
- 9. Subject must have a vertex corrected distance sphero-cylindrical refraction in the range such that appropriate spherical lens powers are available for correction in both eyes. The spherical lens powers available in this study are:

- a. -1.00 to -6.00 (in 0.25D steps)
- 10. Best corrected monocular distance visual acuity must be 20/20<sup>-3</sup> or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

#### **Exclusion Criteria following Screening**

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Be currently using any ocular medications or have any ocular infection of any type.
- 3. By self-report, have any ocular or systemic disease, allergies, or infection, or use medications that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise the study endpoints. See section 9.1 for additional details regarding systemic medications.
- 4. Have previously participated in a contact lens, contact lens package, or lens care related clinical trial.
- 5. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild, or sibling of the employee or their spouse) of the clinical site.

## **Exclusion Criteria at Baseline Evaluation**

The subject must not:

- 6. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings or other corneal, eyelid, or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including significant blepharitis, entropion, ectropion, ptosis, chalazia, recurrent styes, pterygium, significant dry eye disease, history of recurrent corneal erosions, aphakia, corneal distortion, herpetic keratitis).
- 7. Have a history of strabismus or amblyopia.
- 8. Have fluctuations in vision due to clinically significant dry eye or other ocular or systemic conditions.
- 9. Have had or have planned (within the study period) any ocular or intraocular surgery or procedures (e.g., PRK, LASIK, IPL, blepharoplasty, etc.)

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials. Potential study subjects should preferably have a recent history of a comprehensive eye exam, at the investigator's discretion.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This is a 3-visit, multi-site, bilateral, dispensing, non-randomized, uncontrolled, unmasked, single arm study. Subjects will be fitted bilaterally with the same study lenses (one treatment) and dispensed for approximately 2 weeks of wear (two 1-week wear periods). At Visit 1, subjects will be fitted into the study lenses and dispensed for approximately 1 week. At Visit 2 (Follow up #1), additional lenses will be dispensed for another 1-week wearing period. Visit 3 will be the final follow up (#2) and final (exit) evaluation.

At the conclusion of the study, subjects will not have access to the study lenses but will be advised to continue care with their eye care provider (ECP) and discuss contact lens options with them directly.

#### 4.2. Study Design Rationale

Single arm study designs are well-established study designs in which subjects are exposed to a single treatment for the duration of the study. This design is cost effective and efficient when the performance of the treatment is known, and the primary objective of the study is not efficacy related. This design was selected because it most closely simulates real world contact lens fitting experience for subjects, providing an opportunity to measure

commitment to lens wear after a typical contact lens fit and follow-up period. A potential limitation of this design is that it is single arm (uncontrolled), and potential clinical or statistical significance will be limited to the specific treatment and not a general experience of new wearers across various lens brands and their commitment to contact lenses.

#### 4.3. Enrollment Target and Study Duration

This study will have an enrollment target of approximately 40 subjects, and it is estimated that approximately 30 subjects will complete the study. The study will be conducted at up to 5 clinical sites, where the enrollment target for each site will be approximately 8 subjects. A subject will be considered enrolled upon signing of the informed consent/assent form.

The study enrollment period is approximately 8 weeks. Once enrolled, subjects will be in the study for about 2 weeks, making the total study duration about 10 weeks from the first subject first visit (FSFV) to last subject last visit (LSLV). Subjects who are discontinued prior to the final evaluation may be replaced at the discretion of the study sponsor. The investigation will end at the time that the study data is hard locked.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

This study is non-randomized and uncontrolled with the study lenses worn bilaterally in a single arm design.

The following must have occurred prior to lens fitting:

- Informed consent must have been obtained and where applicable assent must have been obtained.
- The subject must have met all eligibility criteria.
- The subject's screening and baseline information must have been collected.

When dispensing test articles, the following should be followed to maintain the Test Article Accountability Log:

Investigator or designee will pull the appropriate test articles from the study supply. All test articles that
are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be
recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 5.2. Masking

This study will be an open label trial. Subjects will be aware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product.

#### 5.3. Procedures for Maintaining and Breaking the Masking

Not Applicable.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test 1 |
|----------------------|--------------------------------|
| Test Article Form | Soft contact lens |
| Design / Description | AO1D (ACUVUE OASYS® 1-DAY with |

| | Test 1 |
|---|---|
| | HydraLuxe™ TECHNOLOGY) |
| Manufacturer | Johnson & Johnson Vision Care, Inc. |
| Packaging Form | Blister packaging in sterile packing solution |
| Packaging Solution | Optimized Borate Buffer (OBB) solution |
| Lens Material | senofilcon A (C3) |
| Sphere Powers (DS) | -1.00 to -6.00 in 0.25 steps |
| Nominal Base Curve (mm) | 8.5 |
| Nominal Lens Diameter (mm) | 14.3 |
| Dk (Fatt method, boundary corrected, edge corrected, ×10 <sup>-11</sup> [cm <sup>2</sup> /sec] [ml O <sub>2</sub> /ml × mm Hg] at 35°C) | 103 |
| Wear Modality in Current Study | Daily wear |
| Replacement Frequency | Daily disposable |

The estimated total number of study lenses that will be required is 1,440. At least 305 lenses per SKU will be made available based on the following factors: sample size, bilateral wear, daily replacement, 2-week dispensing duration, number of sites, safety margin of 1.5X, and US distribution model for the range of lenses -1.00 through -6.00.

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Non-Preserved Rewetting Drops / Saline / Multi-purpose Contact Lens Solution | | |
|---|---|---|---|
| Solution | Single use Eye-Cept® | LacriPure | Biotrue Multipurpose solution |
| Name/Description | Rewetting Drops | Saline Solution | |
| Manufacturer | Optics Laboratory | Menicon | Bausch and Lomb |
| Preservative | None | None | polyaminopropyl biguanide, |
| | | | polyquaternium, and alexidine |

Lens cases and fluorescein strips (either 0.6 mg or 1.0 mg) will be supplied for use as needed.

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the investigator and/or the sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blister packages as the primary packaging and placed into plastic bags as secondary packaging. Sample labels for the primary and secondary packaging are shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions and <u>separate</u> from the <u>site's</u> other related products.

#### 6.6. Collection and Storage of Samples

Used lenses will not be collected as part of the study procedures. When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with enough study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- What was returned to the Investigator unused, including expired or malfunctioning product.
- The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1<br>Screening, Baseline,<br>Treatment 1 | Visit 2<br>Treatment 1 Follow-<br>up 1 | Visit 3<br>Treatment 1 Follow-<br>up 2 |
|---|---|---|---|
| Time Point | Day 0 | 7 ± 1 day following<br>Visit 1 | 7 ± 1 day following<br>Visit 2 |
| Estimated Visit Duration | 4 hours | 2 hours | 2 hours |
| Statement of Informed Consent | X | | |
| Children's Assent (if applicable) | x | | 1 |
| Parent or Legal Guardian<br>Statement of Informed Consent<br>(if applicable) | x | | |
| Demographics | X | | |
| Medical History/Concomitant<br>Medications | x | X | X |
| Eligibility Following Screening | x | | |
| Confidence & Motivation Questionnaire | X | X | x |
| Entrance Visual Acuity | X | X | X |
| Palpebral aperture height (PAH) | X | | |
| Horizontal Visible Iris Diameter<br>(HVID) | х | | |
| Hand dominance | x | | |
| Hand size (Hand length, palm<br>width) | x | | |
| Subjective Sphero-Cylindrical<br>Refraction and best-corrected VA | х | | Х |
| Slit Lamp Biomicroscopy | X | X | x |
| Eligibility Following Baseline<br>Evaluation | x | | |
| Lens Selection | x | | |
| Lens Insertion & Removal<br>Training | x | | |
| Lens Insertion & Removal (timed) | x | х | Х |
| I&R learning session (timed) | x | | |
| Over Refraction and Visual<br>Acuity (if necessary) | X | X | |
| Lens Power Modification (if applicable) | Х | х | |
| Subject Reported Ocular<br>Symptoms | х | x | Х |
| Post Fit Questionnaires | X | | |
| General Fit Assessment | x | X | X |
| Exit Snellen Distance Visual<br>Acuity | x | x | х |
| Dispense Patient Instruction Guide (New wearer contact lens education) | х | | |
| Dispense Test Article | X | X | |
| Lens wear time | | X | X |
| Follow-up Questionnaire | | X | x |

| Visit Information | Visit 1<br>Screening, Baseline,<br>Treatment 1 | Visit 2<br>Treatment 1 Follow-<br>up 1 | Visit 3<br>Treatment 1 Follow-<br>up 2 |
|---|---|---|---|
| Time Point | Day 0 | 7 ± 1 day following<br>Visit 1 | 7 ± 1 day following<br>Visit 2 |
| Estimated Visit Duration | 4 hours | 2 hours | 2 hours |
| Commitment to Lens wear (Exit Interview) | | | x<br>(at Exit Evaluation) |
| Study Completion | | | X |

## 7.2. Detailed Study Procedures

## VISIT 1

The subjects will present to Visit 1 wearing their habitual spectacles or uncorrected.

| | Visit 1: Screening | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.1 | Statement of Informed<br>Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. | |
| | | Note: The subject must be provided a signed copy of this document. | |
| 1.2 | Children's Assent &<br>Parent/Legal guardian<br>Informed Consent (if<br>applicable) | Each minor subject must read (or be read to) and sign the Children's Assent (Information and Assent Form). The parent or legal guardian of the minor must also read, understand, and sign the Statement of Informed Consent (Parental Permission Form and Authorization to Use and Disclose Medical Information). Note: The subject and parent/guardian must be provided a signed copy of these documents. | |
| 1.3 | Demographics | Record the subject's year of birth, age, gender, race and ethnicity. | |
| 1.4 | Medical History and<br>Concomitant<br>Medications | Record the subject's medical history and concomitant medications. | - |
| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" or "N/A" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If the subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms do not need to be completed as part of Final Evaluation. | |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Confidence &<br>Motivation Questionnaire | Subject will complete the baseline Confidence & Motivation Questionnaire directly. |
| 1.7 | Entrance Visual Acuity | Record the distance Snellen visual acuity (OD, OS) to the nearest letter with their habitual spectacles or unaided. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.8 | Palpebral Aperture Height (PAH) | While seated, the subject will direct their gaze straight ahead (primary gaze) and focus on a distant object (e.g., 20/40 letter). Instruct the subject to keep their eyes open naturally (blink as needed). 1. The investigator will measure the palpebral aperture height (PAH) using a mm ruler in the right and left eye. Measurement in mm and to one decimal place. (e.g., 0.0 mm). Note: Minimal illumination should be used as to not cause the subject to 'squint.' If light must be used, allow the subject to adapt to the light for at least one minute. Palpebral aperture height (PAH): vertical distance (blue arrow) between upper and lower eyelid through the center of the pupil. |
| 1.9 | Horizontal Visible Iris<br>Diameter (HVID) | While seated, the subject will direct their gaze straight ahead (primary gaze) and focus on a distant object (e.g., 20/40 letter). Instruct the subject to keep their eyes open naturally (blink as needed). 1. The investigator will measure the Horizontal Visible Iris Diameter (HVID) using a mm ruler in the right and left eye. Hold the millimeter scale across the horizontal meridian. Read the measurement from the |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| | | place. Range 10.0 – 14.0 mm. Average is 11.6. Note: Minimal illumination should be used as to not cause the subject to 'squint.' If light must be used, allow the subject to adapt to the light for at least one minute. The subject's and examiner's eye level should be at the same level. |
| 1.10 | Hand dominance | Horizontal visible iris diameter (HVID): horizontal distance (red arrow) from left and right edge of the iris through the <b>center of the pupil</b> . Record hand preference (hand dominance) for the |
| 1.11 | Hand size | subject. A mm ruler or measuring tape will be used to measure the hand length (HL in diagram) and palm width (PW in diagram) of the right and left hand. Measurement in mm and to one decimal place. |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | PW | |
| 1.12 | Subjective Sphero-<br>cylindrical Refraction | Complete subjective spherocylindrical refraction and record the resultant distance visual acuity (OD and OS) to the nearest letter. | A F |
| 1.13 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If any of these slit lamp findings are grade 3 or higher, the subject may not continue at this time, but may return up to one additional time to determine eligibility. If discontinued a final examination must be completed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline | |
| 1.14 | Eligibility after Baseline | may be instilled. All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If the subject is deemed to be ineligible after baseline, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms do not need to be completed as part of Final Evaluation. | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.15 | Lens Selection | Select the contact lens power based on vertex corrected spherical equivalent of the subjects spherocylindrical refraction. |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.16 | Insertion & Removal training | Study investigator or designated staff will train the subject on insertion and removal of lenses, demonstrating how to retrieve the lenses from the package, position the lens on the finger, secure the eyelids, and how to insert and remove the lenses. | Appendix E |
| 1.17 | I&R Learning Session -<br>Start | Enter the time when I&R learning session begins. | |
| 1.18 | Learning Session:<br>Lens Insertion &<br>Removal | While being timed, the subject will insert and remove the study lenses on their own, one at a time. The Investigator or designated staff will support the subject throughout the learning session. Insertion: Using a stopwatch or a Timer App, record how long it takes the subject to insert each lens (one at a time). • Enter total insertion time OD • Enter total insertion time OS Total insertion time OU Note: | |
| | | <ul> <li>Insertion time starts when the subject first attempts to insert the lens (at the approach step) and stops when the lens is placed on eye.</li> <li>If the lens feels uncomfortable and must be removed, the subject may skip to the lens removal step for that eye. The lens should be inspected for damage and replaced if necessary.</li> <li>If the lens is very uncomfortable needs to be removed immediately, the Investigator or designated staff may do so. The lens should be inspected for damage and replaced if necessary. The Investigator or designated staff will re-insert the lens for the subject.</li> </ul> | |
| | | Removal: Using a stopwatch or a Timer App, observe the subject and record how long it takes them to remove each lens (one at a time). • Total removal time OD • Total removal time OS Total removal time OU Note: • Removal time starts when the subject first attempts to remove the lens (at the approach | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | step) and stops when the lens is successfully removed. • Lenses should be discarded after removal. Note: A slit-lamp examination may be performed at any time during the learning session if the subject's eye(s) seems red or irritated. |
| 1.19 | I&R Learning Session -<br>End | Enter the time when I&R learning session ends. • I&R learning session ends after the subject completes the insertion and removal of both right and left lenses (or when the subject or Investigator stops the learning session). I&R learning session – End Total learning session time OU Note: |
| | | <ul> <li>The learning session may end prematurely if the subject wishes to stop.</li> <li>Investigator may end the learning session prematurely if the subject's eye(s) seems red or irritated, and a slit-lamp examination may be done.</li> <li>Ample time (approximately 1 hour) should be allowed for the subject to practice and complete insertion and removal tasks.</li> <li>If the subject does not complete the learning session within a reasonable time, a second (and final) training opportunity may be provided on a separate day. The subject may return on the following day and up to day 7.</li> </ul> |
| 1.20 | Completion of I&R<br>Learning Session | Record in EDC whether the subject completed the I&R learning session (insertion and removal of lenses at least once for each eye). If a patient did not complete the Learning Session and will come back for a second training/learning session, a second baseline, including Medical History and Concomitant Medications update, Entrance VA, and Slit lamp biomicroscopy will be captured. |
| 1.21 | Patient Instruction<br>Guide (PIG) | Record in EDC that the subject was instructed on proper use and care of contact lenses and provided a copy of the Patient Instruction Guide. Encourage the subject to ask questions and clarify information, if necessary. |
| 1.22 | Lens Selection | Provide the subject a new pair of contact lenses. |
| 1.23 | Lens Insertion | The subject or the Investigator will insert the study lenses. Check for lens damage under the slit lamp before proceeding with lens settling. |

| 0. | I now I | Visit 1: Treatment 1 Lens Fitting |
|---|---|---|
| Step | Procedure | Details |
| 1.24 | Lens Settling | Replace damaged lenses if necessary. Allow the study lenses to settle for a minimum of 10 minutes. |
| | | The subject will spend this time experiencing vision. Instruct the subject to look at distance objects, near objects, and experience bright & dim lighting conditions. |
| 1.25 | Subjective Best Sphere<br>Over Refraction | Perform the monocular subjective best sphere refraction over the study lenses with a phoropter, trial lenses, or flipper bars (adopt the maximum plus to maximum visual acuity). Record distance visual acuity to the nearest letter (OD and OS). |
| 1.26 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not Plano. For each power modification, select the adjusted fitting lens power as appropriate and repeat steps 1.23 through 1.26. |
| 1.27 | Subject Reported Ocular | Up to two power modifications are allowed. Subjects will respond to a verbal open-ended |
| OCT 1 | Symptoms | symptoms questionnaire. |
| 1.28 | General Lens Fit Assessment Confidence & | Evaluate lens centration, movement on blink, and push-up test for each eye. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement. edge lift. excessive movement in primary and up gaze. insufficient movement in all three of the following conditions: primary gaze, up gaze, and push-up test. Note: If lens fit is unacceptable for either eye, the subject will be discontinued from the study. The subject will complete the Confidence & |
| 1.29 | Motivation<br>Questionnaire | Motivation Questionnaires directly. |
| 1.30 | Post-Fit Questionnaire | The subject will complete the Post-Fit Questionnaire directly. |
| 1.31 | Exit VA | Record the subject's distance visual acuity, OD and OS, to the nearest letter. |
| 1.32 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity is 20/30 or better OD and OS. • The lens fit is acceptable OD and OS. • Investigator approval. |

| CA | D | Visit 1: Treatment 1 Lens Fitting |
|---|---|---|
| Step | Procedure | Details If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 1.33 | Dispense | The lenses will be dispensed for a 6-8 day wearing period. Subjects will be encouraged to wear the study lenses every day, building up the wearing time if necessary. The lenses will be worn in a daily wear, daily disposable modality. Rewetting drops are permitted if needed. The subject should only use the sponsor supplied lens care products. (Section 6.1) Supply the subject a bottle of contact lens solution or saline for rinsing purposes, if necessary. Instruct subjects to return any unworn lenses to the clinical site. Subjects will be scheduled for their 1-week follow-up visit, ensuring that they wear the study lens to the follow-up visit. Note: Dispense the subject enough lenses to last them to their next scheduled visit, plus an extra pair. If the subject requires additional replacement lenses, instruct them to contact the clinical site for replacement. As much as reasonably possible, any damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. If the PQC is due to foreign matter in the packaging, to the extent possible, this foreign matter must also be returned. The lens will be stored in labeled vial with saline, and clearly |
| 1.34 | Schedule next visit | differentiated from the other worn lenses that will be shipped back to the Sponsor. • The subject may continue to wear their habitual correction (spectacles) when not wearing study contact lenses. Schedule the follow-up visit to occur in 7 ± 1 days |
| | | (counting the day of this visit as day 0, the subject may return on day 6 through 8). Ensure the subject is instructed to wear the study lenses to the follow-up visit. Remind the subject to bring their spectacle correction to the next visit (if applicable). |

## VISIT 2

The subjects must present to Visit 2 wearing the study lenses. If the subject wishes to stop wearing contact lenses (discontinue), proceed to the Final evaluation.

| | | Visit 2: Treatment 1 Follow-Up 1 |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and<br>Concomitant Medications<br>Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| 2.2 | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 2.3 | Wear Compliance | Confirm the subjects wear schedule. |
| 2.4 | Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.5 | Confidence & Motivation | The subject will complete the Confidence & Motivation Questionnaire directly. |
| 2.6 | Follow-Up Questionnaire | The subject will complete the Follow-Up Questionnaire directly. |
| 2.7 | Entrance Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD and OS) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 2.8 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. |
| | | An unacceptable fit is deemed by one of the following criteria: Imbal exposure at primary gaze or with extreme eye movement. dege lift. excessive movement in primary and up gaze. insufficient movement in all three of the following conditions: primary gaze, up gaze, and push-up test. |
| | | Note: if lens fit is unacceptable subject will be discontinued from the study. |
| 2.9 | Wettability<br>Characteristics | Record the white light lens wettability of both lenses. |
| 2.10 | Surface Deposits | Record any front and back surface lens deposits. |
| 2.11 | Lens Removal (timed) | While being timed, the subject will remove the study lenses, one at a time. Lenses will be temporarily stored in a contact lens case with preservative free saline. Removal: Using a stopwatch or a Timer App, observe the subject and record how long it takes for them to remove each |
| | | lens (one at a time). • Total removal time OD • Total removal time OS Total removal time OU |

| | | Visit 2: Treatment 1 Follow-Up 1 |
|---|---|---|
| Step | Procedure | Details |
| | | Note: • Removal time starts when the subject first attempts to remove the lens (at the approach step) and stops when the lens is successfully removed. |
| 2.12 | Slit Lamp Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the subject has a Grade 3 slit lamp finding, it will be recorded as an Adverse Event and the subject will be monitored as per the guidelines given in section 13. If the clearance of the fluorescein needs to be |
| 2.13 | Lens Insertion (timed) | expedited, preservative-free rewetting drops may be instilled. While being timed, the subject will re-insert the study lenses on their own, one at a time. |
| | | Insertion: Using a stopwatch or a Timer App, observe the subject and record how long it takes for them to insert each lens (one at a time). • Enter total insertion time OD • Enter total insertion time OS Total insertion time OU Note: • Insertion time starts when the subject first attempts to insert the lens (at the approach step) and stops when the lens is placed on eye. • You may ask the subject to let you know when the lens is in. |
| 2.14 | Subjective Best Sphere<br>Over Refraction (if<br>applicable) | An over-refraction <i>may</i> be performed at the Investigators discretion. Perform subjective best sphere refraction over the study lenses with a phoropter, trial lenses, or flipper bars OD and OS. Record the best corrected distance visual acuity to the nearest letter (OD and OS). Note: The subject may continue in the study if the |
| | | over-refraction is Plano, at the Investigators discretion. |
| 2.15 | Lens Power Modification<br>(if applicable) | Adjust the lens power if the subject's best sphere over-<br>refraction is not Plano. |
| 2.16 | Subject Reported Ocular | Up to two power modifications are allowed. Subjects will respond to a verbal open-ended |
| 2.17 | Symptoms (if applicable) Exit VA | symptoms questionnaire. Record the subject's distance visual acuity, OD and |
| 4.1/ | LAILVA | OS, to the nearest letter. |

| | | Visit 2: Treatment 1 Follow-Up 1 |
|---|---|---|
| Step | Procedure | Details |
| 2.18 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity is 20/30 or better OD and OS. • The lens fit is acceptable OD and OS. • Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 2.19 | Dispense | The lenses will be dispensed for a 6-8 day wearing period. Subjects will be encouraged to continue to wear the study lenses every day. The lenses will be worn in a daily wear, daily disposable modality. Rewetting drops are permitted if needed. The subject should only use the sponsor supplied lens care products. Instruct subjects to return any unworn lenses to the clinical site. Subjects will be scheduled for their 1-week follow-up visit, ensuring that they wear the study lens to the follow-up visit. Note: Dispense the subject enough lenses to last them to their next scheduled visit, plus an extra pair. If the subject requires additional replacement lenses, instruct them to contact the clinical site for replacement. As much as reasonably possible, any damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. If the PQC is due to foreign matter in the packaging, to the extent possible, this foreign matter must also be returned. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. The subject may continue to wear their habitual correction (spectacles) when not wearing study contact lenses. |
| 2.20 | Schedule next visit | Schedule the follow-up visit to occur in $7 \pm 1$ days (counting the day of this visit as day 0, the subject may return on day 6 through 8). Ensure the subject is instructed to wear the study lenses to the follow-up visit. Remind the subject to bring their spectacle correction to the next visit (if applicable). |

## VISIT 3

The subjects must present to Visit 3 wearing the study lenses. The subject must bring their habitual spectacles to this visit, if necessary. If the subject wishes to stop wearing contact lenses (discontinue), proceed to the Final evaluation.

| | | Visit 3: Treatment 1 Follow-Up 2 |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and<br>Concomitant Medications<br>Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| 3.2 | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 3.3 | Wear Compliance | Confirm the subjects wear schedule. |
| 3.4 | Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 3.5 | Confidence & Motivation | The subject will complete the Confidence & Motivation Questionnaire directly. |
| 3.6 | Follow-Up<br>Questionnaires | The subject will complete the Follow-Up Questionnaire directly. |
| 3.7 | Entrance Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD and OS) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 3.8 | Subjective Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement. edge lift. excessive movement in primary and up gaze. insufficient movement in all three of the following conditions: primary gaze, up gaze, and push-up test. Note: if lens fit is unacceptable subject will be discontinued from the study. |
| 3.9 | Wettability<br>Characteristics | Record the white light lens wettability of both lenses. |
| 3.10 | Surface Deposits | Record any front and back surface lens deposits. |
| 3.11 | Lens Removal (timed) | While being timed, the subject will remove the study lenses, one at a time. Lenses will be temporarily stored in a contact lens case with preservative free saline. Removal: Using a stopwatch or a Timer App, observe the subject and record how long it takes them to remove each lens (one at a time). Total removal time OD |
| | | Total removal time OS Total removal time OU |

| | Visit 3: Treatment 1 Follow-Up 2 | |
|---|---|---|
| Step | Procedure | Details |
| | | Note: Removal time starts when the subject first attempts to remove the lens (at the approach step) and stops when the lens is successfully removed. |
| 3.12 | Lens Insertion (timed) | While being timed, the subject will re-insert the study lenses on their own, one at a time. Insertion: Using a stopwatch or a Timer App, observe the subject and record how long it takes for them to insert each lens (one at a time). • Enter total insertion time OD • Enter total insertion time OS Total insertion time OU Note: • Insertion time starts when the subject first attempts to insert the lens (at the approach step) and stops when the lens is placed on eye. • You may ask the subject to let you know when the lens is in. |
| 3.13 | Lens Removal | The subject or Investigator will remove the study lenses and discard them. |
| 3.14 | Slit Lamp Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the subject has a Grade 3 slit lamp finding, it will be recorded as an Adverse Event and the subject will be monitored as per the guidelines given in section 13. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Commitment to Lens<br>Wear Questionnaire | The subject will complete the commitment to lens wear Questionnaire directly. |
| F.2 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.3 | Exit Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best-corrected distance visual acuity (OD and OS) to the nearest letter. |

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| | | NOTE: This step is not necessary if the subject was exited due to screen failure. |
| F.4 | Exit Slit Lamp<br>Biomicroscopy (for<br>subjects that are<br>discontinued early) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. This step is not necessary if the subject was exited due to screen failure. NOTE: This step is not necessary if the subject was |
| | | exited due to screen failure, or if biomicroscopy was performed as part of the final follow-up visit procedures (i.e., immediately prior to the final evaluation). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected, as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the
  adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Reason for unscheduled visit | Indicate if the <u>only</u> reason for the visit is that the subject requires additional test articles. If the reason is other than resupply of previously dispensed lenses, specify the reason for the visit. |
| U.2 | Chief Complaints (if applicable) | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.3 | Adverse Events and<br>Concomitant<br>Medications Review (if<br>applicable) | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.4 | Entrance VA (if applicable) | Record the entrance distance visual acuity (OD, OS) to the nearest letter. |

| | Unscheduled Visit | | |
|---|---|---|---|
| Step | Procedure | Details | 3- |
| U.5 | Subjective Sphero-<br>cylindrical Refraction (if<br>applicable) | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS). | |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applicable) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. | |
| U.7 | Dispensing (if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, provide additional lenses per the dispensing instructions given in the detailed study procedures. | |
| U.8 | Exit Visual Acuity (if applicable) | Record the subject's exit distance visual acuity (OD, OS) to the nearest letter. | |

NOTE: If the only reason for the unscheduled visit is that the subject requires additional test articles, only the dispensing information needs to be recorded.

#### 7.4. Laboratory Procedures

None.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

#### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- they are eligible.
- have not withdrawn/discontinued from the study for any reason described in section 8.2.
- completed all visits through the final Visit 3.
- If all visits were completed but an additional visit is considered necessary for subject care, follow the requirements for unscheduled visits in section 7.3.

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject withdrawal of consent.
- Subject not compliant to protocol (e.g., subject wearing the lenses overnight).
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events necessitating temporary or permanent discontinuation of study lens wear.
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Subjects who have experienced a symptomatic ocular adverse event necessitating temporary or permanent discontinuation of study lenses.
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject not compliant with study lens wear schedule (e.g., subject doesn't wear study lenses at all between visits).
Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort
or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless
  otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

Additional subjects may be enrolled if a subject discontinues from the study prematurely, at the Sponsor's discretion.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study.

Disallowed medications for this study include: Any ocular (ophthalmic) or systemic medications that may contraindicate contact lens wear or may compromise study endpoints, at the Investigators discretion.

Concomitant therapies that are disallowed include: Any therapy the investigator believes may contraindicate contact lens wear.

#### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film.

A summary of disallowed systemic medications is shown in Table 4. Subjects with an active history of taking these medications will not be allowed to enroll.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Vitamin A analogs | Cystic acne | Isotretinoin |
| Corticosteroids | Various inflammatory conditions such as<br>Rheumatoid Arthritis, inflammatory<br>bowel diseases (Crohn's, Ulcerative<br>Colitis), Systemic Lupus Erythematosus,<br>dermatological conditions (Eczema,<br>Psoriasis), Chronic Uveitis, etc. | Prednisone, dexamethasone, methylprednisolone, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report

deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 5 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 5: Examples of major and minor protocol deviations

| Deviation category | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | Visit attended more than 2 days out of visit window defined in study procedures | Visit attended 2 or fewer days out<br>of visit window defined in study<br>procedures |
| Unanswered PRO questions or surveys | For questionnaires where data is related to a primary endpoint, one or more PRO questions or other pertinent questions are unanswered (i.e., left blank). | For questionnaires where data is related to an exploratory endpoint, one or more PRO questions are unanswered (i.e., left blank). |
| Time for insertion | N/A | Time is not recorded for an I&R session and any data related the exploratory endpoints is missing. |
| Subject wears the lenses on an Extended Wear (EW) schedule | Subject sleeps in study lenses overnight | N/A |

In the case of a major protocol deviation, the decision of whether or not the subject will be excluded from the Per-Protocol analysis population will be made at the time of cohort review.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor will review with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness, or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e., tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also apply and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated."

NOTE: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

NOTE: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear.

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Contact Lens-induced Acute Red Eye (CLARE)
- Any Temporary Loss of > 2 Lines of BCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

NOTE 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.<sup>1</sup>

**Unanticipated Adverse Device Effect (UADE)** – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in section 13.2.2).
- Outcome not recovered or not resolved, recovering, or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.

Actions Taken – none, temporarily discontinued, permanently discontinued, or other.

#### 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's
  daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study, it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.

- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

In the event of a serious/significant adverse event, the Investigator must:

Notify the Sponsor immediately.

- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None.

#### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical analysis will be undertaken by the study biostatistician. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC<sup>6</sup>. Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables, and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics

(n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

#### 14.2. Sample Size Justification

This study was not designed or powered to test any statistical hypotheses, as there was no available data for these endpoints and population. The sample size of 40 subjects to enroll with approximately 30 to complete was based on clinical considerations and operational feasibility to gain more understanding about the new wearers contact lens experience.

#### 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article.

#### **Per-Protocol Population:**

All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification for the exclusion of subjects with protocol deviations from the per-protocol population set will be documented in a memo to file.

#### **Intent-to-Treat (ITT) Population:**

Intention-to-treat population will include all assigned subjects.

#### 14.4. Level of Statistical Significance

Not applicable, there is no planned hypothesis testing for any study endpoints.

#### 14.5. Primary Analysis

The primary analyses will be conducted on the safety population. The primary endpoint will be summarized using counts and percentages. The primary endpoints will be evaluated using the following clinical findings:

Incidence (percentage) of eyes with Grade 3 or 4 slit lamp findings related to the study lenses after 2-week of lens wear.

#### 14.6. Secondary Analysis

Not applicable.

#### 14.7. Exploratory Analysis

The exploratory analyses will be conducted on the Intention-to-Treat population.

The following endpoints will be collected and analyzed separately for each timepoint:

- 1. Commitment to lens wear: Do you want to continue to wear contact lenses after this study?
- 2. Reasons for Discontinuation (if applicable): Which of the following is the main reason why you want to stop wearing contact lenses?
- 3. Insertion Time OU (at the initial fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear).
- 4. Removal time OU (at the initial fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear).
- Confidence (baseline, post fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear).
- 6. Motivation (baseline, post fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear).
- 7. Lens performance (CLUE vision, comfort, and handling scores) at fitting, after approximately 1-week of wear, and after approximately 2-weeks of wear.

In addition, the relationship between endpoints (i.e., CLUE<sup>™</sup> scores, insertion time (OU), and removal time (OU) and human factors will also be investigated both graphically (e.g., via scatterplots) and through a correlation analysis, at fitting and 1-week follow-up.

Anatomical human factors will include palpebral aperture height (PAH), horizontal visible iris diameter (HVID), hand length, palm width, hand dominance and while non-anatomical human factors will include motivation, confidence, and demographics (e.g., gender, age).

#### 14.8. Interim Analysis

Not applicable.

#### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using the Sitero EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis. Data generated from post hoc measurements (e.g., Compositional characteristics of contact lens lipid uptake, Measured tear film protective capability, Measured contact lens surface dehydration rate, etc.) will be collected on specific Microsoft Office Excel format worksheets at the clinical site and at the completion of the analysis transferred to JJVC biostatistician for data analysis in such format.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2020.<sup>1</sup>

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent

- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. To allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 16.4. Data Monitoring Committee (DMC)

Not applicable.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects and their parents/legal guardians will be fully informed of the risks and requirements of the study and, during the study, subjects and their parents/legal guardians will be given any new information that may affect their decision to continue participation. Subjects and their parents/legal guardians will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Subjects will only be enrolled if the subject is / subject's parents/legal guardians are fully able to understand the risks, benefits, and potential adverse events of the study and provide their consent voluntarily, and the subject provides their assent voluntarily.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, according to ISO 14155:2020,¹ and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64th WMA General Assembly 2013² and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with applicable regulatory requirements.

#### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

#### For subjects aged 18 or older

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH GCP<sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

#### For subjects aged 13 to 17

Each subject must give written assent and their parents (legal guardians) must give written consent according to local requirements after the nature of the study has been fully explained. The consent and assent forms must be

signed before performance of any study-related activity. The consent and assent forms that are used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent and assent are in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH GCP<sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject and the parent (legal guardian) the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects and their parents (legal guardians) will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject and parent (legal guardian) will be given sufficient time to read the Information and Assent form and the informed consent form (Parental Permission Form and Authorization to Use and Disclose Medical Information), respectively, and the opportunity to ask questions. After this explanation and before entry into the study, assent and consent should be appropriately recorded by means of the subject's and parent/legal guardian's dated signatures. After having obtained the consent and assent, a copy of the informed consent and assent forms must be given to the subject.

#### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>7</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel, and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, except for Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ISO 14155:2020,¹ guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ISO 14155:2020,¹ and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

There is no plan to publish the outcome of this investigation.

#### 22. REFERENCES

1. ISO 14155:2020: Clinical Investigation of Medical Devices for Human Subjects — Good Clinical Practice. Available at: https://www.iso.org/standard/71690.html

- 2. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects.

  Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 3. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 4. Sulley A, et. al., Retention rates in new contact lens wearers. Eye & Contact Lens 2018.
- 5. Wirth RJ, Edwards MC, Henderson M, Henderson T, Oliveres G, Houts CR. Development of the contact lens user experience: CLUE scales. *Optometry and Vision Science*. 2016;93(8):801-8. https://pubmed.ncbi.nlm.nih.gov/27383257/
- 6. SAS Institute Inc: SAS® 9.4 Statements: Reference, Third Edition. Cary, NC SAS Institute Inc; 2014.
- 7. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)













Confidential







### APPENDIX B: PATIENT INSTRUCTION GUIDE

A patient instruction guide (PIG) will be provided separately

### APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

ACUVUE OASYS® 1-DAY with HydraLuxe™ TECHNOLOGY (AO1D)

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology for ASTIGMATISM

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear



## SYMBOLS KEY

The following symbols may appear on the label or carton:

| SYMBOL | SYMBOL DEFINITION |
|---|---|
| [i] | Consult Instructions for Use |
| | Manufactured by or in |
| M | Date of Manufacture |
| 8 | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterile Using Steam or Dry Heat |
| 2 | Single-Use |
| DIA | Diameter |
| BC | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylinder |
| AXIS | Axis |
| <b>C€</b><br>0086 | Quality System Certification Symbol |
| UV Blocking | UV-Blocking |
| 0 | Fee Paid for Waste Management |
| R <sub>X</sub> Only | CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner |
| ₩ ♦ | Lens Orientation Correct |
| W W | Lens Orientation Incorrect (Lens Inside Out) |

## DESCRIPTION

ACUVUE OASYS® Brand Contact Lenses 1-Day and ACUVUE OASYS® Brand Contact Lenses 1-Day for ASTIGMATISM are soft (hydrophilic) contact lenses made with HydraLuxe™ Technology. They are available as spherical or toric lenses respectively.

These lenses are made of a silicone hydrogel material containing an internal wetting agent, visibility tint, and UV absorbing monomer and are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling.

A benzotriazole UV absorbing monomer is used to block UV radiation. The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

### Lens Properties:

### The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 - 1.12

Refractive Index: 1.42

Light Transmission:
 85% minimum

Surface Character: Hydrophilic

Water Content: 38%

Oxygen Permeability:

#### VALUE METHOD

122 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, non-(ml O<sub>2</sub>/ml x mm Hg) at 35°C edge corrected)

103 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge (ml O<sub>2</sub>/ml x mm Hg) at 35°C corrected)

#### Lens Parameters:

Diameter Range: 12.0 mm to 15.0 mm
Center Thickness: varies with power
Base Curve Range: 7.85 mm to 10.00 mm
Spherical Power Range: -20.00D to +20.00D
Cylinder Power Range: -0.25D to -10.00D
Axis Range: 2.5° to 180°

## AVAILABLE LENS PARAMETERS

ACUVUE OASYS® Brand 1-Day with HydraLuxe™ Technology are hemispherical shells of the following dimensions:

Diameter: 14.3 mm

Center Thickness: 0.085 mm to 0.221 mm (varies with power)

Base Curve: 8.5 mm, 9.0 mm

Powers: -0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in 0.50D increments) +0.50D to +6.00D (in 0.25D increments) +6.50D to +8.00D (in 0.50D increments)

ACUVUE OASYS® Brand 1-Day with HydraLuxe™ Technology for ASTIGMATISM are hemitoric shells of the following dimensions:

Diameter: 14.3 mm

**Center Thickness:** 0.075 mm to 0.172 mm (varies with power)

Base Curve: 8.5 mm

**Powers:** +0.00D to -6.00D (in 0.25D increments)

Cylinders: -0.75D, -1.25D, -1.75D, -2.25D\*

Axis: 10° to 180° in 10° increments

\*-2.25D cylinder is available in 10°, 20°, 70°, 80°, 90°, 100°, 110°,

160°, 170°, 180° axes only.

+0.25D to +4.00D (in 0.25D increments)

-6.50D to -9.00D (in 0.50D increments)

Cylinders: -0.75D, -1.25D, -1.75D

Axis: 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

### TRANSMITTANCE CURVES

ACUVUE OASYS® 1-Day with HydraLuxe™ Technology (senofilcon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



<sup>\*</sup> The data was obtained from measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-9.00D lens, 0.075 mm center thickness).

Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21

<sup>2</sup>Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

## **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays onto the retina.

The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

## INDICATIONS (USES)

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™
Technology are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astigmatism.

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.

These lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

## CONTRAINDICATIONS (REASONS NOT TO USE)

# DO NOT USE these contact lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye.
- Any eye disease, injury or abnormality that affects the cornea, conjunctiva, or eyelids.
- Severe insufficiency of lacrimal secretion (dry eye).

- Corneal hypoesthesia (reduced corneal sensitivity).
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use of contact lens solutions (i.e., rewetting drops) that contain chemicals or preservatives (such as mercury, Thimerosal, etc.) to which some people may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

### **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION; IF THE PATIENT EXPERIENCES:

- Eye Discomfort,
- Excessive Tearing,
- Vision Changes,
- Loss of Vision,
- Eye Redness,
- Or Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY RE-MOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

 When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Clinical studies have shown that the risk of serious adverse reactions is increased when lenses are worn overnight, and that the risk of ulcerative keratitis is greater for
extended wear contact lens users than for daily wear users.3

- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.
- The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

#### Specific Instructions for Use and Warnings:

Water Activity

#### Instructions for Use

Do not expose contact lenses to water while wearing them.

#### WARNING:

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

### **PRECAUTIONS**

### Special Precautions for Eye Care Professionals:

• Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

<sup>&</sup>lt;sup>3</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

- The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.
- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Fluorescein, a yellow dye, should not be used while the lenses are
  on the eyes. The lenses absorb this dye and become discolored.
   Whenever fluorescein is used in eyes, the eyes should be flushed
  with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove the lenses immediately if the eyes become red or irritated.

## Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

#### **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the "Patient Instruction Guide" for the prescribed

wearing schedule and those prescribed by the Eye Care Professional.

- Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container unless specifically indicated for that use. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernails.

#### **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens." The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.
- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.
- Always discard lenses worn as prescribed by the Eye Care Professional.

#### **Lens Care Precautions:**

 The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

#### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed. Depending on the severity, this could include the use of lubricating drops that are indicated for use with soft contact lenses or the temporary discontinuance of contact lens wear while such medication is being used.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

### **ADVERSE REACTIONS**

# The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- . There may be the potential for some temporary impairment due to

peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis; some of which are clinically acceptable in low amounts.

- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows, or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be instructed NOT to use a new lens as self-treatment for the problem.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

#### **GENERAL FITTING GUIDELINES**

#### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- · Motivation to wear lenses
- · Ability to follow instructions regarding lens wear care
- General health
- · Ability to adequately handle and care for the lenses
- . Ability to understand the risk and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

#### **B. Pre-fitting Examination**

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

#### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than  $\pm 4.00D$ ,

#### D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.

- ACUVUE OASYS® 1-Day: 8.5 mm/14.3 mm
- ACUVUE OASYS® 1-Day for ASTIGMATISM: 8.5 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

#### 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

#### 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink, and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

#### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

### E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |

| Example 2 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see dispensing and follow up information in **PATIENT MANAGEMENT**).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing ACUVUE OASYS® 1-Day for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

### A. How to Determine Lens Cylinder and Axis Orientation

#### 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position – there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.



You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

#### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

#### 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift", measure or estimate the "drift", then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

#### **B. Final Lens Power**

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

#### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx  $> \pm 4.00$ D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq \pm 4.00$ D, vertex compensation is not necessary.

#### 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq$  0.50D from the refractive cylinder.

#### 3. Case Examples

#### Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20

O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx Prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

#### Example 2

Manifest (spectacle) refraction: O.D. -3.00D / -1.00D x 90° 20/20 O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power, cylinder power, and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

#### Right Eye

The orientation mark on the right lens rotates left from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx Prescribed: O.D. -3.00D / -0.75D x 100°

#### Left Eye

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position.

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx Prescribed: O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow-up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot meet state driver's licensing requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

#### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision and straight ahead and upward gaze that monovision contact lenses provide.

#### **B. Eye Selection**

#### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1: Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

#### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

### C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require corrective lenses on

both eyes.

#### Examples:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the GENERAL FITTING GUIDELINES for base curve selection described in this Package Insert.

Case history and standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under

conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

### D. Other Suggestions

The success of the monovision technique may be further improved by having the patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation.
   Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### PATIENT MANAGEMENT

#### **Dispensing Visit**

Each sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. To remove the lens from the container, peel back the foil seal, place a finger on the lens, and slide the lens up the side of the bowl of the lens package until it is free of the container.

- · Evaluate the physical fit and visual acuity of the lens on each eye.
- Teach the patient how to apply and remove his or her lenses.
- Explain daily disposable lens wear and schedule a follow-up examination.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

### Follow-Up Examinations

Follow-up care (necessary to ensure continued successful contact lens wear) should include routine periodic progress examinations, management of specific problems, if any, and a review with the patient of the wear schedule, daily disposable modality, and proper lens handling procedures.

Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis):

- 1. One week from the initial lens dispensing to patient
- 2. One month post-dispensing
- 3. Every three to six months thereafter

**NOTE:** Preferably, at the follow-up visits, lenses should be worn for at least six hours.

#### Recommended Procedures for Follow-up Visits:

- 1. Solicit and record patient's symptoms, if any.
- 2. Measure visual acuity monocularly and binocularly at distance and near with the contact lenses.
- Perform an over-refraction at distance and near to check for residual refractive error.
- With the biomicroscope, judge the lens fitting characteristics (as described in the **GENERAL FITTING GUIDELINES**) and evaluate the lens surface for deposits and damage.
- 5. Following lens removal, examine the cornea and conjunctiva with the biomicroscope and fluorescein (unless contraindicated).
  - The presence of vertical corneal striae in the posterior central cornea and/or corneal neovascularization is indicative of excessive corneal edema.
  - The presence of corneal staining and/or limbal-conjunctival hyperemia can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear and/or a poorly fitting lens.
  - Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.
- Periodically perform keratometry and spectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are abnormal, use professional judgment to alleviate the problem and restore the eye to optimal conditions. If

the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

### WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to overwear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

The maximum suggested wearing time for these lenses is:

| Day | Hours |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

### REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

### LENS CARE DIRECTIONS

When lenses are prescribed for daily disposable wear, the Eye Care Professional should provide the patient with appropriate and adequate warnings and instructions for daily disposable lens wear at the time they are dispensed.

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have spare lenses or spectacles available.

#### **Basic Instructions**

- Always wash, rinse, and dry hands before handling contact lenses.
- Do not use saliva or anything other than the recommended solutions for lubricating or rewetting lenses. Do not put lenses in the mouth.
- Eye Care Professionals may recommend a lubricating/rewetting solution which can be used to wet (lubricate) lenses while they are being worn to make them more comfortable.

#### Care for a Sticking (Non-Moving) Lens

If the lens sticks (stops moving), the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should immediately consult the Eye Care Professional.

### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

### **HOW SUPPLIED**

Each UV-blocking sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. The plastic package is marked with the following:

- ACUVUE OASYS® 1-Day: base curve, power, diameter, lot number, and expiration date
- ACUVUE OASYS® 1-Day for ASTIGMATISM: base curve, power, diameter, cylinder, axis, lot number, and expiration date

## REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

Tel: 1-800-843-2020

www.acuvue.com



©Johnson & Johnson Vision Care Companies 2016 In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed in USA.

Revision date: 09/16

Revision number: AO-03-16-13

ACUVUE OASYS® and HydraLuxe™ are Trademarks of the Johnson & Johnson Vision Care Companies

### APPENDIX D:

| • | LENS FITTING CHARACTERISTICS | |
|---|----------------------------------------------------|-------------|
| • | SUBJECT REPORTED OCULAR SYMPTOMS | |
| • | FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCED | OURE |
| • | DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRA | CTIVE ERROR |
| • | BIOMICROSCOPY SCALE | |
| • | DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION | 1 |
| • | PATIENT REPORTED OUTCOMES | |
| • | WHITE LIGHT LENS SURFACE WETTABILITY | |



Johnson & Johnson Vision Care, Inc. Lens Fitting Characteristics Title: **Document Type: Document Number:** Revision Number: 6

Johnson & Johnson Vision Care, Inc. Lens Fitting Characteristics Title: Document Type: **Document Number:** Revision Number: 6

Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Lens Fitting Characteristics Title: Document Type: Document Number: Revision Number: 6

Johnson & Johnson Vision Care, Inc. Lens Fitting Characteristics

| Title: | Lens Fitting Characteristics | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number</b> | : | Revision Number: 6 |



Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Lens Fitting Characteristics Title: **Document Type:** 

Document Number: Revision Number: 6





**Clinical Study Protocol** Johnson & Johnson Vision Care, Inc. Subject Reported Ocular Symptoms/Problems Title: Document Type: **Document Number:** Revision Number: 4



Johnson & Johnson Vision Care, Inc. Front and Back Surface Lens Deposit Grading Procedure

Title: **Document Type: Document Number: Revision Number: 4** 

Johnson & Johnson Vision Care, Inc. Front and Back Surface Lens Deposit Grading Procedure

Title: **Document Type: Document Number: Revision Number: 4** 

Johnson & Johnson Vision Care, Inc. Front and Back Surface Lens Deposit Grading Procedure Title: Document Type: **Document Number:** Revision Number: 4



Johnson & Johnson Vision Care, Inc.

| Title: | Front and Back Surface Lens Deposit Grading Proce |
|----------------|---------------------------------------------------|
| Document Type: | |

Document Type:

Document Number: 4

Revision Number: 4




Johnson & Johnson Vision Care, Inc. Determination of Distance Spherocylindrical Refractive Error

Title: **Document Type: Document Number: Revision Number: 5** 











Title: **Biomicroscopy Scale Document Type: Document Number:** Revision Number: 10

Page 1 of 5

Title: **Biomicroscopy Scale Document Type: Document Number:** Revision Number: 10

| Title: | Biomicroscopy Scale | |
|-----------------------|---------------------|---------------------|
| <b>Document Type:</b> | | |
| Document Number: | 7 | Revision Number: 10 |



Page 3 of 5

Title: **Biomicroscopy Scale Document Type: Document Number:** Revision Number: 10

Title: Biomicroscopy Scale

Document Type:

Document Number: Revision Number: 10



Johnson & Johnson Vision Care, Inc. Distance and Near Snellen Visual Acuity Evaluation Title: Document Type: Document Number: **Revision Number: 5** 

Johnson & Johnson Vision Care, Inc. tance and Near Snellen Visual Acuity Evaluation

| Γitle: | Distance and Near | r Snellen Visual Acuity Ev | valuation |
|----------------|-------------------|----------------------------|-----------|
| Document Type: | | | |



Johnson & Johnson Vision Care, Inc. Distance and Near Snellen Visual Acuity Evaluation

**Document Type: Document Number: Revision Number: 5** 

Title:

Johnson & Johnson Vision Care, Inc. Distance and Near Snellen Visual Acuity Evaluation

| Title: | | ar Snellen Visual Acuity Evaluation | |
|---|---|---|---|
| <b>Document Type:</b> | | | |
| <b>Document Number</b> | : | _ | Revision Number: 5 |





| TO LA | Johnson & Johnson Vision Care, Inc. | | |
|---|---|---|---|
| Title: | Patient Reported Outcomes | | |
| Document Type:<br>Document Number: | | Revision Number: | 3 |
| | | • | |



| Title: | White Light Lens Surface Wettability | | |
|---|---|---|---|
| Document Type: Document Number: | - | Revision Number: | 2 |
| Document Number. | | _ 1.01131011111111111111111111111111 | |
| , | | | |
| | | | _ |
| | | | _ |

APPENDIX E: WORK AID: INSERTION AND REMOVAL TRAINING GUIDE











CR-6565, v 2.0 JJVC 



CR-6565, v 2.0 JJVC 



CR-6565, v 2.0 JJVC CONFIDENTIAL






CR-6565, v 2.0 (14) 





CR-6565, v 2.0 JJVC 



9

APPENDIX F: GUIDELINES FOR COVID-19 RISK MITIGATION

| Litle: | Guidelines for CC | OVID-19 Risk Mitigation | |
|---|---|---|---|
| Document Type: | | | |
| Document Number: | | | Revision Number: 6 |

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for clinical study sites participating in Johnson & Johnson Vision Care (JJVC) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVC) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. This Work Instruction will be reviewed and updated as needed.

As of May 2023, the World Health Organization (WHO) declared an end to COVID-19 as a public health emergency. The Centers for Disease Control and Prevention (CDC) also updated its Interim Infection Prevention and Control Recommendations for Healthcare Personnel During the Coronavirus Disease 2019 (COVID-19) Pandemic in May 2023. References for regulations and industry guidelines can be found in the Resource Links section below.

Evaluation of sites outside of the United States (OUS) will be performed on a country-by-country basis subject to local health authority guidance. If the OUS site resides in a country requiring greater than standard of care practices to prevent the spread of COVID-19 in an optometric setting, this guidance can be applied for the JJVC clinical study at that site.

This work instruction can also be utilized for sites within the United States if changes in government recommendations occur or based on the preference of the clinical site, or investigator.

#### 3.0 DEFINITIONS

American Academy of Optometry (AAO): The American Academy of Optometry is an organization of optometrists based in Orlando, Florida. Its goal is to maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometrists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometric Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 Doctors of Optometry (O.D.), optometric professionals, and optometry students. Doctor of Optometry take a leading role in patient care with respect to eye and vision care, as well as general health and well-being. As primary health care providers, Doctor of Optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a federation of state, student, and armed forces optometric associations. Through these affiliations, the AOA serves members consisting of optometrists, students of optometry, paraoptometric assistants and technicians. The AOA and its affiliates work to provide the public with quality vision and eye care.

Centers for Disease Control and Prevention (CDC): The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federal agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** Current outbreak of respiratory disease caused by a novel coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 6

Clinical Study: Voluntary research studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing treatments. May also be called clinical trials, studies, research, trials, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

Clinical Operations Manager (COM): The Johnson & Johnson Vision Care (JJVC) individual responsible for the overall management of a clinical trial.

**Monitor:** An individual designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulatory requirements.

**Medical Safety Officer (MSO):** Physician who has primary accountability in their product portfolio for product health and safety, and who serves as an independent medical voice for patient safety.

Safety Management Team (SMT): A cross-functional, collaborative team responsible for review, assessment and evaluation of medical safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JJVC is providing recommendations for study-related management in the event of disruption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of participants and site staff. If, at any time, a participant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study participants and study personnel:

#### 4.1 Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavirus infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with health care professionals during the procedures and assessments (since the investigator must make the measurements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the virus, even if they do not have symptoms.
- Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment
  due to COVID-19 restrictions. In this event, all assessments that can be conducted virtually will be
  completed by the investigator to determine the best course of treatment for the subject, including
  an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during participation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 6

To help minimize the above potential risks, JJVC recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JJVC will provide the following study specific documents with language pertaining to COVID-19 risks:

#### 4.1.1 Informed Consent:

Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed Consent document:

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

It is important to note that this study will be conducted, at least in part, during the COVID-19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is particularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-term serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on current knowledge from the Centers for Disease Control and Prevention (CDC), those at high-risk for severe illness from COVID-19 include older adults and people with underlying medical conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conformance to guidance from the CDC, local health departments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

If you are found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be permitted to continue in-office study follow-up visits, but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

#### 4.1.2 COVID-19 Risk Control Checklist (Attachment-B):

Will include COVID-19 risk control methods that are required by a site to conduct JJVC clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principal Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

#### 4.1.3 Protocol Compliance Investigator(s) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and governmental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JJVC pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

#### 4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 6

#### 5.0 GUIDANCE FOR REMOTE SUBJECT VISITS

Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-up visits.

Subjects may be delayed in being seen for study follow up visit(s), for example due to COVID-19 control measures or due to the subject's concerns or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:

| Procedure | Details |
|---|---|
| Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and<br>Compliance | Record the average wearing time (including number of hours per day during weekdays and weekends, and number of days per week). Confirm compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-report. For example, the subjects will be asked the time of the day the subject typically puts on the study lenses in the morning and takes off in the evening, the number of days per week lenses were worn, and the number of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all unused lenses to the clinic at the last visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case report forms should capture specific information regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURING PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including Optometry Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Every effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be performed to the extent possible remotely/virtually or delayed until such time that on-site


uidelines for COVID 10 Disk Mitigation

| Title: | Guidelines for CO | OVID-19 Risk Mitigation | |
|---|---|---|---|
| Document Type: | | | |
| Document Number | | | Revision Number: 6 |

visits can be resumed in order to continue participant monitoring in accordance with the protocol where possible. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible.

Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Interruptions of test article wear or discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19related" in the case report form (CRF).

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible monitor to discuss initial plans for study intervention and follow-up. The monitor will notify the Safety Management Team of any subject(s) that have reported "COVID-19", "Asymptomatic COVID-19", "COVID-19 Exposure", or "Suspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study report.

#### 6.1 **Monitoring Visits**

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing limitations during this COVID-19 pandemic, all routine operations related to clinical trials should be well-documented and archived as part of standard process. When conditions permit, all parties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently informed.

#### 6.1.1 Study Site Initiation:

During the period that this Work Instruction is in effect, Site Initiation Meetings and training of study site staff may be conducted remotely. The JJVC study team will conduct training via Skype. Zoom, Microsoft Teams or similar software as well as utilize online training materials, as applicable. Study site training will be documented utilizing Site Initiation Report per Study Site Initiation

On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

#### 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits may be kept to a minimum and include only those tasks that the CRA cannot perform remotely (e.g., source document verification, test article reconciliation, etc.).

To ensure data integrity during the conduct of all JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 6

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

### 6.1.3 Study Site Closure:

During the period that this Work Instruction is in effect, the duration of the Study Site Closure Visit may be limited to tasks that the CRA cannot perform remotely (e.g., source document verification, test article final reconciliation and return, etc.).


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 6

### Attachment A: Study Site Correspondence

MONTH DD, YYYY

Re: COVID-19 Mitigation Plan, << CR-xxxx/protocol title>>

Dear << Principal Investigator>> and Study Team,

Coronavirus (COVID-19) has impacted several communities and business activities over the past several years. While we work toward the successful conduct of clinical studies, our commitment continues to be the safety of patients, healthcare professionals, and to our communities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Vision Care company sponsored clinical trial(s) you are currently working on or considering participation within.

### **Protocol:**

Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

#### Protocol Signature Page:

 Will include a statement indicating the Principal Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

#### **Informed Consent:**

 Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed consent document.

#### **COVID-19 Risk Control Checklist for Clinical Studies:**

 Will include COVID-19 risk control measures that are required to ensure the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication about potential challenges you may foresee as the result of the current COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study correspondence.


| Title: | Guidennes for Co | OVID-19 KISK MINGAHON | | |
|---|---|---|---|---|
| Document Type: | | | | |
| Document Number: | | | Revision | Number: 6 |

#### Attachment B: COVID-19 Risk Control Checklist

Study Number Site Number Principal Investigator (PI) Name

The following risk control operational measures are to be implemented in order to mitigate the risks of contracting COVID-19 illness by patients and/or staff participating in Johnson & Johnson Vision Care (JJVC) clinical studies. Any local regulations, industry guidelines and COVID-19 policy at the institution/clinic should be followed in addition to this checklist.

| PI Initials | General Site Safety Planning Measures |
|---|---|
| | Signage within site describing Risk Control methods |
| | Social Distancing practices throughout site (waiting rooms, lobby, exam rooms, etc.) |
| | Training on patient flow and physical distancing in waiting room |
| | Establish longer time frame between patient appointments to reduce persons in the site |
| | Staff should receive job-specific training on PPE and demonstrate competency with selection and proper use of PPE and wear at all times during interactions with subjects (e.g., putting on and removing without self-contamination) |

| PI Initials | Site Staff Daily Safety Measures |
|---|---|
| | As part of routine practice, site staff should regularly monitor themselves for fever and symptoms |
| | of COVID-19, including temperature checks |
| | Any staff member (including non-study clinic staff and Investigators) showing signs of being sick |
| | or testing positive for COVID-19 must not be permitted to work on activity that may expose study |
| | related staff and subject and the Sponsor shall be informed |
| | NOTE: Inform JJVC in 24 hours of any COVID-19 cases and all potential exposure during |
| | the clinical study. |
| | Ensure that all staff wear a mask |
| | Gloves should be worn if there is physical direct patient contact and changed between each patient |
| | Have staff thoroughly wash hands for at least 20 seconds or use an alcohol-based hand sanitizer |
| | when they arrive, before and after each patient, before eating and after using the bathroom. |
| | Cleaning and disinfection procedures for exam rooms and instruments or equipment between |
| | patients with gloves. |
| | Cleaning and disinfection procedures for commonly touched surfaces (doors, chairs, computers, |
| | phones, etc.) with gloves. |

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to entering the site about fever and respiratory illness and whether |
| | they or a family member have had contact with another person with confirmed COVID-19 in the |
| | past 14 days. Patients exhibiting signs of being sick should be rescheduled when their symptoms |
| | resolve. Patients who have had close contact with someone with confirmed or suspected COVID- |
| | 19 infection should contact the site to report exposure. |

| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| Document Type: | | |
| Document Number: | | Revision Number: 6 |

| PI Initials | Patients Entering the site: |
|---|---|
| | All patients and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise |
| | seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned regularly. |

I certify that I have read and agree to implement all the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Vision Care studies. I agree to the disclosure of potential risks due to COVID-19. If any of the risk mitigation precautions change during the course of the study, I will contact Johnson & Johnson. I understand the possible risks of COVID-19 transmission if our facility's measures are not aligned with the above.

Principal Investigator Signature and Date


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 6

#### RESOURCE LINKS

 WHO chief declares end to COVID-19 as a global health emergency: https://news.un.org/en/story/2023/05/1136367

### **US Resource Links**

- CDC Interim Infection Prevention and Control Recommendations for Healthcare Personnel During the Coronavirus Disease 2019 (COVID-19) Pandemic <a href="https://www.cdc.gov/coronavirus/2019-ncov/hcp/infection-control-recommendations.html">https://www.cdc.gov/coronavirus/2019-ncov/hcp/infection-control-recommendations.html</a>
- OSHA Protecting Workers: Guidance on Mitigating and Preventing the Spread of COVID-19 in the Workplace: https://www.osha.gov/coronavirus/safework
- CDC Training for Healthcare Professionals: <a href="https://www.cdc.gov/coronavirus/2019-ncov/hcp/training.html">https://www.cdc.gov/coronavirus/2019-ncov/hcp/training.html</a>
- I&R Training ACUVUE® LensAssist: <a href="https://www.acuvue.com/lensassist">https://www.acuvue.com/lensassist</a>
- American Optometric Association COVID-19 latest updates: <a href="https://www.aoa.org/covid-19/covid-19-latest-updates">https://www.aoa.org/covid-19/covid-19-latest-updates</a>

#### **OUS Resource Links**

- Hong Kong
  - Updates on local regulations: <a href="https://www.coronavirus.gov.hk/eng/index.html">https://www.coronavirus.gov.hk/eng/index.html</a>
- England
  - NHS Updates and Guidance for Optical Settings: <a href="https://www.england.nhs.uk/coronavirus/publication/updates-and-guidance-for-optical-settings/">https://www.england.nhs.uk/coronavirus/publication/updates-and-guidance-for-optical-settings/</a>
- United Kingdom
  - The College of Optometrists primary eye care COVID-19 guidance: <a href="https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html">https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html</a>
  - NHS advice about COVID-19, including symptoms, testing, vaccination and staying at home: https://www.nhs.uk/conditions/coronavirus-covid-19/
  - Canada
    - COVID-19 for health professionals: Infection prevention and control: https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavirus-infection/health-professionals/infection-prevention-control.html
  - Australia
    - Optometry Australia: Infection control guidelines and advice <u>Infection control guidelines and</u> advice - Optometry Australia

### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6565 Evaluation of Acuvue Oasys 1-Day contact lenses in new wearers

Version and Date: 2.0 12 March 2024

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020,¹ the Declaration of Helsinki,² United States (US) Code of Federal Regulations (CFR),³ and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. I, as the Principal Investigator, am responsible for ensuring that all clinical site personnel, including Sub-Investigators, adhere to all regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| _ | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | · · · · · · | |
| | Institution/Site Name | |
| | institution/site Name | |
| | Institution/Site Address | |